CLINICAL TRIAL: NCT02001857
Title: Effect of TachoSil® on Incidence of Symptomatic and Radiographic Lymphoceles After Extended Pelvic Lymph Node Dissection in Prostate and Bladder Cancer.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EC/2013/472; 2013-000782-36 (EudraCT Number)
Record Dates: First submitted 2013-10-28; First posted 2013-12-05 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Prostate or Bladder Cancer
Keywords: patients,; undergoing; pelvic; lymph; node; dissection.
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TachoSil (Experimental): TachoSil
  Interventions: Drug: 1 TachoSil hemostatic sponge (9,5 cm x 4,8 cm) placed on each side on the external iliac artery.
- No TachoSil (No Intervention): No TachoSil

INTERVENTIONS:
Drug: 1 TachoSil hemostatic sponge (9,5 cm x 4,8 cm) placed on each side on the external iliac artery. — at the end of surgery
  Arms: TachoSil

SUMMARY:
Pelvic lymph node dissection (PLND) is the most accurate staging tool to determine lymph node involvement in prostate and bladder cancer. The main complication of PLND is development of a lymphocele, which can cause symptoms including lower abdominal pain, leg or penile/scrotal edema, bladder outlet obstruction, deep venous thrombosis or infection/sepsis. The incidence of radiographic (asymptomatic) and symptomatic lymphoceles following PLND varies between 12,6-63% and 1,6-33% respectively. Medicated sponges such as Tachosil® are indicated in surgery for improvement of haemostasis and to promote tissue sealing. They could reduce lymphocele development by increased tissue sealing, due to a mechanical effect of the sponge itself and a lymphostatic effect of the included thrombin and fibrinogen. Our goal is to prospectively assess the lymphostatic effect of Tachosil(r) in patients undergoing transperitoneal PLND with or without radical prostatectomy or PLND with bladder cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Diagnosis of prostate cancer or bladder cancer on pathology
* Undergoing transperitoneal pelvic lymph node dissection.

Exclusion Criteria:

* Previous pelvic surgery or irradiation.
* Any type of clotting disorder.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-09; Primary Completion 2017-02 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
development of a radiographic lymphocele on abdominal ultrasonography | at week 1 post-surgery
volume of radiographic lymphoceles | at week 1 post-surgery
duration of postoperative drainage catheter | Daily during standard postoperative care until removal of the catheter, with an expected average of 1 day.
volume produced by postoperative drainage catheter (lymphorrhea) | Daily during standard postoperative care until removal of the drain, with an expected average of 1 day.
time between operation and first flatus, first peristalsis, first passing of stool and removal of gastrostomy tube (signs of ileus recuperation). | Daily during standard postoperative care up to date of first flatus, first peristalsis, first passing of stool and removal of gastrostomy tube (signs of ileus recuperation), with an expected average of 1 day.
  specific for bladder cancer
development of a radiographic lymphocele on abdominal ultrasonography | at week 4 post-surgery
volume of radiographic lymphoceles | at week 4 post-surgery

SECONDARY OUTCOMES:
development of a symptomatic lymphocele. | at week 1 post-surgery
decrease in serum hemoglobin on the first postoperative day | at week 1 post-surgery
duration of hospital stay | at week 1 post-surgery
total cost | at week 1 post-surgery
  Total cost includes: surgical procedure, hospitalization and possible complications up to the first month post-surgery.
development of a symptomatic lymphocele. | at week 4 post-surgery
decrease in serum hemoglobin on the first postoperative day | at week 4 post-surgery
duration of hospital stay | at week 4 post-surgery
total cost | at week 4 post-surgery
  Total cost includes: surgical procedure, hospitalization and possible complications up to the first month post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas Lumen, MD, PhD, FEBU, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium